CLINICAL TRIAL: NCT07182591
Title: A Phase 1, Open-label, Multicenter, First-in-Human Trial of DS5361b in Participants With Advanced Solid Tumors
Brief Title: A Study of DS5361b in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS5361-061
Record Dates: First submitted 2025-08-27; First posted 2025-09-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor
Keywords: First-in-Human; Advanced Solid Tumors
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Monotherapy (Dose Escalation) (Experimental): Participants will receive DS5361b at escalating doses.
  Interventions: Drug: DS5361b
- Part 2: Combination Therapy (Dose Escalation) (Experimental): Participants will receive DS5361b at escalating doses in combination with Pembrolizumab.
  Interventions: Drug: DS5361b; Drug: Pembrolizumab
- Part 3: Combination Therapy (Dose Expansion) (Experimental): Participants will receive DS5361b in combination with Pembrolizumab at the recommended dose for expansion (RDE).
  Interventions: Drug: DS5361b; Drug: Pembrolizumab

INTERVENTIONS:
Drug: DS5361b — Dose Escalation Part: DS5361b will be administered at escalating doses to determine the RDE.
  Dose Expansion Part: DS5361b will be administered at RDE.
Drug: Pembrolizumab — Dose Escalation Part: Pembrolizumab will be administered at a standard dose.
  Dose Expansion Part: Pembrolizumab will be administered at a standard dose.
  Other Names: Keytruda®
  Arms: Part 2: Combination Therapy (Dose Escalation); Part 3: Combination Therapy (Dose Expansion)

SUMMARY:
This study aims to assess the safety, tolerability, and preliminary efficacy and to determine the MTD of DS5361b in monotherapy and combination with pembrolizumab in participants with advanced or metastatic solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

The clinical site will screen for the full inclusion criteria per protocol.

1. Adults ≥18 years of age at the time the ICF is signed (Please follow local regulatory requirements if the legal age of consent for trial participation is >18 years old).
2. Has histologically- or cytologically documented recurrent, metastatic, or unresectable solid tumors that are refractory to or intolerable with standard treatment or for which no standard treatment is available (For Part 1 and Part 2 only).
3. Participants need to have documented TMB or MSI status using a validated or approved genomic test as per applicable regulations prior to Cycle 1 Day 1. In Part 1 and Part 2, participants need to have documented TMB-H and/or MSI-H status. In Part 3, participants need to have documented TMB-H status.
4. Has measurable disease based on local CT/MRI imaging as assessment by the investigator using RECIST v1.1.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
6. Has adequate organ and bone marrow function as assessed by local laboratory within 14 days prior to initiation of trial intervention.
7. For HNSCC participants only: have documented results from local testing of HPV for oropharyngeal cancer. If HPV status has previously been tested using this procedure, no retesting is required.

   Dose Expansion (Part 3) Only:
8. Has histologically or cytologically confirmed, Stage IV NSCLC without actionable gene alteration.

   * No prior systemic therapy.
   * Participants with PD-L1 TPS ≥1%.
9. Has histologically or cytologically confirmed recurrent or metastatic HNSCC that is considered incurable by local therapies.

   * No prior systemic therapy administered in the recurrent or metastatic setting.
   * Participants with PD-L1 CPS ≥1.

Key Exclusion Criteria:

1. Has spinal cord compression or clinically active central nervous system metastases.
2. Has a history of leptomeningeal carcinomatosis.
3. Uncontrolled or significant cardiovascular disease.
4. Any of the following within the past 6 months prior to enrollment: cerebrovascular accident, transient ischemic attack, or other arterial thromboembolic event.
5. Has a history of (noninfectious) interstitial lung disease (ILD)/pneumonitis that required corticosteroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out.
6. Clinically severe pulmonary compromise (ie, requiring any supplemental oxygen).
7. Has any evidence of severe or uncontrolled systemic diseases.
8. Has active or uncontrolled HBV infection. Hepatitis B SCR testing is required.
9. Has active or uncontrolled HCV infection. Hepatitis C SCR testing is required.
10. For the dose escalation phase (Part 1 and Part 2), has HIV infection. For the dose expansion part (Part 3), has active or uncontrolled HIV infection.
11. Prior organ transplantation, including allogeneic stem cell transplantation.
12. Has an active, known, or suspected autoimmune disease.
13. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the trial intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2030-03-18 (Estimated); Study Completion 2030-12-03 (Estimated)

PRIMARY OUTCOMES:
Part 1 and 2: Number of participants with Dose-Limiting Toxicities (DLTs) | Cycle 1: Day 1 up to Day 21 (each cycle is 21 days)
  A DLT is defined as any Treatment Emergent Adverse Event (TEAE) not attributable to disease or disease-related processes, environmental factors, unrelated trauma, etc, that occurs during the DLT evaluation period (Day 1 to the end of Cycle 1) and is Grade ≥3.
Part 1, 2, and 3: Number of Participants Experiencing a Treatment Emergent Adverse Event (TEAE) | From Screening up to approximately 5 years
  TEAEs are defined as those Adverse Events (AEs) with start or worsening date during the on-treatment period (from the first dose date of trial intervention to 30 days after the last dose date of trial intervention).
Part 3 Only: Objective Response Rate (ORR) Following the Administration of DS5361b at RDE(s) in Combination with Pembrolizumab | From first dose up to approximately 5 years
  ORR is defined as the proportion of participants with a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), as assessed by investigator per RECIST v1.1.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of DS5361b | Cycle 1: Day 1, Day 15 (each cycle is 21 days)
Time to Reach Maximum Plasma Concentration (Tmax) of DS5361b | Cycle 1: Day 1, Day 15 (each cycle is 21 days)
Area Under the Plasma Concentration-time Curve up to the Last Quantifiable Time (AUClast) of DS5361b | Cycle 1: Day 1 (each cycle is 21 days)
Trough Plasma Concentration (Ctrough) of DS5361b | Cycle 1: Day 15 (each cycle is 21 days)
Part 1 and 2: Objective Response Rate (ORR) Following the Administration of DS5361b Alone and in Combination with Pembrolizumab | From first dose up to approximately 5 years
  ORR is defined as the proportion of participants with a BOR of confirmed CR or PR, as assessed by investigator per RECIST v1.1.
Disease Control Rate (DCR) Following Administration of DS5361b Alone and in Combination with Pembrolizumab | From first dose up to approximately 5 years
  DCR is defined as the proportion of participants who achieved a BOR of confirmed CR, confirmed PR, or stable disease as assessed by investigator per RECIST v1.1.
Duration of Response (DoR) Following Administration of DS5361b Alone and in Combination with Pembrolizumab | From first dose up to approximately 5 years
  DoR is defined as the time (in months) from date of initial response (CR or PR) to the earlier date of the first objective documentation of radiographic disease progression or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Research Site, Sarasota, Florida
  - Brown University School of Medicine, Providence, Rhode Island
  - Research Site, Irving, Texas
  - Research Site, San Antonio, Texas
- Research Site, Kashiwa, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/